CLINICAL TRIAL: NCT02568410
Title: Platelets as Regulators of Inflammation and Tissue Injury After Cardiac Surgery
Brief Title: Platelets as Regulators of Inflammation in Cardiac Surgery
Acronym: PRICS
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00064249
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2018-06

CONDITIONS: Systemic Inflammatory Response Syndrome; Acute Kidney Injury
Keywords: Mast Cells; Blood Platelets; cardiac surgical procedures
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, DNA, Platelet RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CABG on CPB: Patients undergoing elective coronary artery bypass grafting using cardiopulmonary bypass. No study interventions beyond the standard clinical practice for these surgeries at Duke University Medical Center. No study drug administration.
  Interventions: Procedure: coronary artery bypass grafting using cardiopulmonary bypass

INTERVENTIONS:
Procedure: coronary artery bypass grafting using cardiopulmonary bypass — no study intervention. Study cohort will undergo coronary artery bypass grafting using cardiopulmonary bypass according to standard practices at DUMC

SUMMARY:
Platelets are increasingly recognized as a potent and ubiquitously present source of inflammatory activation. Importantly, antiplatelet therapy has been shown to significantly reduce major adverse events such as renal injury in cardiac surgery patients. However, in current practice, concerns of excessive bleeding-not platelet activation and thrombosis-shape clinical decisions.

The investigators have recently seen, that a significant drop in platelet numbers following cardiac surgery is associated with increased mortality and risk of acute kidney injury. The investigators hypothesize that such thrombocytopenia is a result of excessive perioperative platelet activation and resultant release of inflammatory and tissue injurious signals by activated platelets. Platelet activation will be characterized during and after cardiac surgery and examine its correlation with inflammatory responses and perioperative end-organ injury.

DETAILED DESCRIPTION:
Distant organ injury is a frequent consequence of cardiovascular surgery involving cardio-pulmonary bypass. Acute kidney injury (AKI), the most common complication, occurs in 30%-40% of cardiac surgery patients and, even with moderate damage, significantly increases mortality and healthcare costs. Although organ injury has been linked to inflammation, the mechanisms that initiate and propagate these events remain poorly defined. As the median age and medical complexity of cardiac patients increases, the challenge - and opportunity - to improve organ protection lies in identifying modifiable targets.

The investigators preliminary work provides primary evidence that activated platelets play a novel role in the initiation of tissue injurious and inflammatory responses at the microvascular interface. As such, platelets aggregate in close proximity to perivascular mast cells, a cell type that can rapidly launch powerful inflammatory responses through release of preformed effectors. Platelet activation alone is sufficient to stimulate these mast cells in vitro while, conversely, pharmacological inhibition of platelets reduce mast cell-dependent inflammation and end organ injury after rat circulatory arrest.

Based on compelling experimental data and evidence of human relevance, the investigators have formed our central hypothesis that platelet activation is an important trigger of inflammatory and tissue injurious responses after cardiopulmonary bypass through stimulation of perivascular mast cells. The objective is to define the pathophysiologic relevance of the platelet/mast cell interaction to end organ injury, and to identify targets for novel strategies of organ protection in cardiac surgery patients.

Specific Aim: Define platelet activation as a risk factor for end organ injury in cardiac surgery patients.

The investigators preliminary data strongly suggest that thrombocytopenia after cardiac surgery is linked to AKI and increased mortality. In a prospective study of 100 patients undergoing coronary artery bypass graft (CAGB) surgery, the investigators will define platelet activation and consumption as the likely cause of this thrombocytopenia, and establish the association between platelet activation in general with markers of mast cell activation, systemic inflammation, and AKI.

Approach:

The objective of this aim is to investigate the link between perioperative platelet activation, systemic inflammatory responses, and adverse end organ outcomes.

The investigators will perform a prospective observational study of 100 patients to investigate the link between perioperative platelet activation, systemic inflammatory responses, and end organ injury following cardiac surgery. Patient inclusion criteria for this study will be based on the results from our retrospective study of 4201 patients undergoing CABG surgery on CPB. Here, the investigators identified a significant incidence of thrombocytopenia and an association between thrombocytopenia and increased risk for developing postoperative AKI. Consequently, the proposed study is designed to determine whether postoperative platelet activation contributes to a systemic inflammatory response and, hence, has a causative effect on end organ injury.

Sample collection and processing: 15 mL of venous blood will be drawn into ACD buffer before incision and at 10 minutes, and 6, 24, 48, and 72 hours after separation from cardiopulmonary bypass (CPB).

Measurements: The investigators will analyze serum platelet markers by enzyme-linked immunosorbent assay (ELISA) and the characteristic changes in membrane protein expression by multicolor Fluorescence-activated cell sorting (FACS). Corresponding platelet counts will be determined at each time point. Aspirin medication is given until the day of surgery and again starting on postoperative day 2 as standard of care. Because aspirin resistance may influence our outcomes, the investigators will measure 11-dehydrothromboxane B2 urine levels. Ensuing subgroup analysis will establish the relevance of aspirin resistance to our observations. Systemic inflammation will be examined by determining the plasma cytokine levels by ELISA. As an additional arm of investigation the investigators will collect patient DNA and platelet RNA to further examine the genomic characteristics and platelet gene expression profiles associated with an enhanced platelet activation during surgery. This data will inform further studies in personalized identification of risk factors for patients undergoing cardiac surgery.

Primary outcome: AKI is a clinically relevant manifestation of end organ injury and will serve as our primary outcome. With an incidence of 30%-40% following cardiac surgery, the investigators expect to observe a sufficient number of cases of AKI to allow adequate statistical analysis. The investigators will define AKI according to Kidney Disease: Improving Global Outcomes (KDIGO) criteria and record AKI using both the proposed stages and the change in serum creatinine values from 3 days before to 10 days after the surgery date.

Secondary outcomes: The investigators will measure cytokine expression and platelet activation as secondary outcomes. Further, the investigators will also collect established measures of clinical outcome such as hospital length of stay, ICU length of stay, duration of postoperative mechanical ventilation, and major adverse cardiac events (MACE) defined as all-cause mortality, emergent revascularization, atrial fibrillation, stroke, and non-fatal myocardial infarction.

Patient characteristics and numbers, power-analysis, and patient Data collection: Variables will be recorded from patient files: 1) preoperatively: age, gender, race, Society of Thoracic Surgery risk factors, EUROScore, date of consent, and preoperative drugs; 2) intraoperatively: number of coronary artery bypass grafts, duration of cardio-pulmonary bypass, duration of aortic cross clamp, cumulative dose of heparin administered, blood products, and cumulative dose of sympathomimetic and vasopressor drugs; 3) postoperatively: timing of complications, cause and timing of death, hospital and ICU length of stay, duration of postoperative mechanical ventilation, dose of inotropic or vasoactive support. Plate-let count and creatinine levels, as well as anti-platelet therapy will be recorded from 3 days be-fore to 10 days after the surgery.

Expected Outcomes. In this Aim, the investigators expect to provide new insights into the origins of systemic inflammation and end organ injury following cardiac surgery. Our preliminary data indicate that postoperative thrombopenia is associated with AKI and mortality. The investigators expect to demonstrate that such thrombocytopenia occurs in a setting of ongoing platelet activation and is associated with systemic inflammation and, ultimately, end organ injury. Together, these investigations will lay the foundation for novel organ protection strategies in cardiac surgery.

Statistical analysis. Descriptive comparisons will be made by using Kruskal-Wallis test or chi-square test, as appropriate. Univariable and multivariable linear or logistic regression analyses will be applied, as appropriate, to evaluate the association between the primary and secondary outcomes and pre-, intra-, and postoperative variables. R2 for linear regression analyses, odds ratios, and the corresponding 95% confidence limits for logistic regression analyses will be re-ported.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing elective CABG procedures

Exclusion Criteria:

* patients with a history of:

  * renal injury (creatinine > 1.5 mg/dL)
  * hepatic insufficiency (liver function tests > 1.5 times the upper limit of normal),
  * severe pulmonary insufficiency (requiring home oxygen therapy),
  * EF < 20%,
  * IABP use preoperatively,
  * liver, heart, or lung transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective coronary artery bypass grafting
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2015-10; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | 30 days
  AKI according to KDIGO criteria

SECONDARY OUTCOMES:
systemic inflammatory response activation, as measured by serum TNFa levels | perioperative
  serum measurement of inflammatory markers
systemic inflammatory response activation, as measured by serum IL8 levels | perioperative
  serum measurement of inflammatory markers
systemic inflammatory response activation, as measured by serum Chymase levels | perioperative
  serum measurement of inflammatory markers
systemic inflammatory response activation, as measured by serum IL6 levels | perioperative
  serum measurement of inflammatory markers
platelet activation, as measured by p-selection levels | perioperative
  p-selectin, serum platelet factor 4
platelet activation, as measured by serum platelet factor 4 levels | perioperative
  p-selectin, serum platelet factor 4
hospital length of stay | 30-days
Intensive care unit length of stay | 30-day
major adverse cardiac events | 30-day
  all-cause mortality, emergent revascularization, atrial fibrillation, stroke, and non-fatal myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: jorn karhausen, md, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States